CLINICAL TRIAL: NCT03062748
Title: Predicting Cardiometabolic Risk in Mild-to-Moderate Obstructive Sleep Apnea: Inflammation vs. Apnea/Hypopnea Index
Status: Enrolling by invitation | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Alexandros Vgontzas, Professor, Milton S. Hershey Medical Center
Other Study IDs: 5218
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to compare the relative contribution of systemic inflammation vs. Obstructive Sleep Apnea (OSA) severity (as measured by Apnea Hypopnea Index) in predicting cardiovascular and metabolic aberrations associated with mild-to-moderate obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate OSA (5≤ AHI <30)
* BMI ≤ 45
* Age ≥ 18
* Men & Women

Exclusion Criteria:

* AHI ≥ 30
* BMI >45
* Current use of steroids or anti-inflammatory medication
* Diagnosis of insulin dependent diabetes
* Diagnosis of autoimmune disorder
* Shiftwork
* Current use of CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected OS who are being seen at the Sleep Research and Treatment Center.
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence of the metabolic syndrome | baseline
  At least 3 of the following 5 risk factors must be met in order to have the metabolic syndrome:
  1. Elevated waist measurement (≥102 cm for men or ≥89 cm for women)
  2. Elevated triglycerides (≥150 mg/dL or use of medication)
  3. Low HDL cholesterol (<50 mg/dL for women or <40 mg/dL for men or use of medication)
  4. Elevated blood pressure (≥130 mmHg systolic or ≥ 85 mmHg diastolic or use of medication)
  5. Elevated fasting blood sugar (≥100 mg/dL or use of medication)
  Source: https://www.nhlbi.nih.gov/health/health-topics/topics/ms
Obstructive Sleep Apnea | baseline
  AHI from one night polysomnography
Markers of systemic inflammation | baseline
  CRP, IL-6, TNFa

SECONDARY OUTCOMES:
Heart rate variability | baseline
  from polysomnography
Subjective measure of sleepiness | baseline
  Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No